CLINICAL TRIAL: NCT03407092
Title: Thrombectomy In ANdalucia Using Aspiration (TRIANA)
Acronym: TRIANA
Status: Completed | Type: Observational
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Collaborators: Andaluz Health Service (Other Government)
Responsible Party: Principal Investigator, Alejandro González, Principal Investigator, Hospitales Universitarios Virgen del Rocío
Other Study IDs: PI-0374-2017
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stentriever Cohort
  Interventions: Other: Stentriever Cohort
- ADAPT cohort
  Interventions: Other: ADAPT cohort

INTERVENTIONS:
Other: ADAPT cohort — Thrombectomy with distal aspiration technique
  Groups: ADAPT cohort
Other: Stentriever Cohort — Thrombectomy with stent retriever
  Groups: Stentriever Cohort

SUMMARY:
This study aims to compare the efficacy and safety of ADAPT vs Stentriever techique in a multicenter stroke cohort of patients.

DETAILED DESCRIPTION:
In Andalusia, current data show that the mortality rate from stroke is 50% higher than in Spain as a whole. Endovascular therapy has revolutionized the treatment of acute stroke and could improve these high mortality rates. The investigators propose to take the great advance that the thrombectomy has given to the community of Andalusia in which there are more limited resources with several strategies such as the implementation of strict protocols of inclusion through a common registry, use of cheaper equipment (aspiration vs stent-retrievers)

The objective of the TRIANA trial is thus to:

1. Demonstrate that the use of thrombectomy systems with direct aspiration first pass technique (ADAPT ) using the new large-bore 6F SOFIA Plus catheter (MicroVention, Inc., a wholly owned subsidiary of Terumo Corporation) is equal in safety and efficacy to the results of thrombectomy with stent retriever.

2) The use of mechanical aspiration systems would lead to a decrease in cost per procedure, shortening the duration of treatment and decrease the rate of embolism to new territory.

3) Identify futile recanalization blood biomarkers that will allow the investigators in the future to treat only those patients who will benefit from the most adequate reperfusion treatment.

The design is an observational, prospective and multicentric study of patients with acute ischemic stroke of anterior circulation and less than 8 hours of evolution treated with neurointerventionist rescue techniques to study safety, effectiveness, costs of the intervention and duration (puncture-recanalization) of the thrombectomy system with aspiration with Sofia Plus in comparison with the stent retrievers system.

1. To evaluate the safety and effectiveness of thrombectomy with manual mechanical aspiration with Sofia Plus under clinical practice conditions.
2. Determine if the duration (puncture-recanalization) of thrombectomy with aspiration is less than that of stents retrievers; And if the number of embolisms distal to new vascular territories decreases with aspiration.
3. To estimate the cost savings by procedure in the treatment of ischemic stroke and to analyze the efficiency (cost effectiveness) of thrombectomy with aspiration.

ELIGIBILITY:
Inclusion Criteria:

* Subject experiencing an acute ischemic stroke in which imaging demonstrates a vascular occlusion located in the distal internal carotid artery (ICA) through the distal middle cerebral artery (MCA).
* Subjects in which the aspiration technique is used for at least the first two thrombectomy passes per occluded vessel.
* Subjects older than 18 years old.
* Subjects with a prestroke modified Rankin scale of 0-2 and presenting with an NIHSS of 2-30.
* Subjects that the operator feels may be treated with endovascular therapy.
* Subjects in which computed tomography (CT)/Magnetic Resonance Imaging (MRI) demonstrates an infarct size of less than 70cc on MRI or Alberta Stroke Program Early CT (ASPECTS) score overall of 6 or better.
* Subjects in which groin puncture can be obtained within 6 hours of symptom onset (with or without Total Plasminogen Activator administration). In those Patients of more than 8 hours or awake stroke or of unknown onset should be individualized the treatment and must exist area of penumbra in CT perfusion.
* Subjects who have consented in accordance with local Institutional Review Board requirements.

Exclusion Criteria:

* Absence of large vessel occlusion on neuroimaging.
* Platelet count < 100 x 10³ cells/mm³ or known platelet dysfunction.
* Contraindication to CT and/or MRI (i.e., due to contrast allergy or prior implant that precludes MRI imaging).
* Previously documented contrast allergy that is not amenable to medical treatment.
* Women who are pregnant or breastfeeding at time of intervention.
* Evidence of brain hemorrhage on CT and/or MRI at presenting hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with ischemic stroke in which imaging demonstrates a vascular occlusion located in the distal internal carotid artery (ICA) through the distal middle cerebral artery (MCA) who require endovascular reperfusion.
Sampling Method: Non-Probability Sample
Enrollment: 532 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
modified rankin scale (mRs) at 90 days | 90 days
  Is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
  Score Description: The scale runs from 0-6, running from perfect health without symptoms to death.
  0 No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead

SECONDARY OUTCOMES:
Symptomatic Intracranial bleeding | during admission
Haemorrhagic tranformation | during admission
  Haemorrhagic tranformation in control computed tomography after thrombectomy.
Thrombolysis in cerebral infarction (TICI) scale | Up to 24 hours after endovascular reperfusion
  It´s a tool for determining the response of thrombolytic/thrombectomy therapy for ischaemic stroke. In neurointerventional radiology it is commonly used for patients post endovascular revascularisation. Like most therapy response grading systems, it predicts prognosis.
  Classification
  The description is based on the angiographic appearances of the treated occluded vessel and the distal branches:
  Grade 0: no perfusion Grade 1: penetration with minimal perfusion Grade 2: partial perfusion Grade 2A: only partial filling (less than two-thirds) of the entire vascular territory is visualized Grade 2B: complete filling of all of the expected vascular territory is visualized but the filling is slower than normal Grade 3: complete perfusion

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro González, Md, PhD, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Spain

IPD SHARING:
Plan to Share IPD: No